CLINICAL TRIAL: NCT02349620
Title: Platelet-rich Factot in Implant Dentistry
Brief Title: Effect of Platelet-rich Factor on Implant Stability and Bone Resorption in the Lower Posterior Mandible
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reza Tabrizi (Other)
Responsible Party: Sponsor-Investigator, Reza Tabrizi, Assistant professor of shahid beheshti university of medical sciences, Shiraz University of Medical Sciences
Organization: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2014-10-05; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Osseointegrated Dental Implantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A:partialy edutolus patients (Active Comparator): In this group surface treated implant with PRF will be inserted.Immediately after the surgery the implant stability will be measure with the Osstell mentor to verify the resonance frequency analysis (RFA), using the smart peg type 1, then stability will be measured every 2 weeks up to 3 months .Bone height will be measured in mesial and distal side immediately after placement and in months 3 and 6 with Intra Oral Peri Apical xray (IOPA x-ray)
  Interventions: Biological: PRF
- B: partialy edutolus patients (Placebo Comparator): In this group implant with out PRF will be inserted.Immediately after the surgery the implant stability will be measured with the Osstell mentor to verify the resonance frequence analysis (RFA ), using the smartpeg type 1, then stability will be measured every 2 weeks up to 3 months. Bone height was measured in mesial and distal side immediately after placement and in months 3 and 6 with IOPA xray

INTERVENTIONS:
Biological: PRF — implant stability was measured by RFA and implant resorption was measured by IOPA after surface treatment by PRF
  Arms: A:partialy edutolus patients

SUMMARY:
The main objective of this clinical trial study is to consider the effect of Platelet-Rich-Factor (PRF) on implant stability and marginal bone resorption around dental implants.

DETAILED DESCRIPTION:
Dental implants were placed in 30 subjects who have 1 or 2 missing teeth in both side of posterior mandible. Implants with a length of 11.5 and a diameter of 4.5 mm will be inserted in both sides. In one side PRF will be instilled after surface treatment with PRF before implant placement, while no PRF was added in other side to serve as control group. All implants will be followed with stability measurement by means of resonance frequency analysis at baseline, and every two weeks up to 3 months. Bone height was measured on medial & distal side on standardized IOPA x-rays.

ELIGIBILITY:
Inclusion Criteria:

* patients who have 1 or 2 missing teeth in both side of posterior mandible

  * adequate bone quantity and quality at the implant site
  * the implant sites with at least 3 months of healing after extraction,
  * patients well motivated for implant therapy and maintaining good oral hygiene
  * the implant sites with width and length to installation of an implant of 4.5 mm x 11.5 mm.
  * Patients who gave written informed consent

Exclusion Criteria:

* • medically compromised or patients taking any immunosuppressive drugs which may complicate the treatment outcome

  * infection around the implant site
  * history of bruxism/parafunctional habits
  * patients with history of any bleeding disorder or on anti-coagulant therapy.
  * pregnant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
implant loss | 6 months
  During the osseointegration, if the implant lose his stability and if the patient have pain, the implant will be removed and the implant will be considered lost

SECONDARY OUTCOMES:
ISQ analysis | 3 months
  Since the implant installation, the implant stability will be measure with the Osstell, that will return a number between 0 and 100. This represents the Implant Stability Quotient (ISQ). The difference between the ISQ results will be the secondary outcome measure
bone height (mm) | 6 months
  Since the implant insertion , bone height was measured in mesial and distal side on standardized IOPA x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Reza Tabrizi, DMD, Study Chair — Shiraz University of Medical Sciences; Touba karagah, DMD, Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Shiraz university of medical sciences, Shiraz, Fars, Iran